CLINICAL TRIAL: NCT05864625
Title: Comparison of Hemodynamic Stability During Anesthesia Using Remimazolam and Sevoflurane in Patients Undergoing Minimally Invasive Aortic Valve Replacement Surgery : A Prospective Randomized Controlled Study
Brief Title: Comparison of Hemodynamic Stability During Anesthesia Using Remimazolam and Sevoflurane in Minimally Invasive AVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Assistant professor for fund, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 05-2023-105
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Aortic Valve Stenosis; Remimazolam
Keywords: Aortic Valve Stenosis; Remimazolam
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Long-Term Synaptic Depression; Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam (Experimental): Induction dose of 6 mg/kg/h of remimazolam with remifentanil TCI 1~4 nanogram/mL are injected together. When patient loses consciousness, rocuronium 0.8 mg/kg is given and endotracheal intubation is performed after confirming that TOF count is less than one. Anesthesia is maintained by using remimazolam dose of 1mg/kg/h~2mg/kg/h with remifentanil to maintain optimal depth of anesthesia, which will checked by Sedline value between 25 to 50.
  Interventions: Drug: Remimazolam besylate
- Propofol/sevoflurane (Active Comparator): 1% propofol 1-2mg/kg is injected with remifentanil TCI 1~4, and when patient loses consciousness, sevoflurane is started and rocuronium 0.8mg/kg is given. After confirming that TOF count is less than one, intubation is performed and anesthesia is maintained with sevoflurane and remifentanil to keep the Sedline value between 25 and 50.
  Interventions: Drug: Propofol/ Sevoflurane

INTERVENTIONS:
Drug: Remimazolam besylate — During induction, patients allocated to the remimazolam group will receive remimazolam 6mg/kg/h with remifentanil TCI 1~4 nanogram/mL. After patient loses consciousness, anesthesia will be maintained with remimazolam 1-2mg/kg/h combied with remifetanil.
  Other Names: Remimazolam besylate, Byfavo Inj., Hana Pharm Col, Ltd., Seoul, Korea
  Arms: Remimazolam
Drug: Propofol/ Sevoflurane — During induction, patients allocated to the P/S group will receive propofol 1% 1-2mg/kg with remifentanil TCI 1~4 nanogram/mL. After patient loses consciousness, anesthesia will be maintained with sevoflurane and remifentanil.
  Other Names: Fresofol 1% TM, Fresenius
  Arms: Propofol/sevoflurane

SUMMARY:
Anesthetic agents can cause hypotension, and be especially dangerous in patients with severe aortic stenosis, which can lead to even circulatory collapse. Remimazolam is known for its hemodynamic stability compared to propofol. This study is designed to compare effects of remimazolam vs. sevoflurane anesthesia on intraoperative hemodynamics in patients with severe aortic valve stenosis.

DETAILED DESCRIPTION:
Anesthetic agents can cause hypotension due to reduced cardiac contractility and vasodilation. This can be especially dangerous in patients with severe aortic stenosis, which can lead to even circulatory collapse in extreme cases. Remimazolam is a relatively new anesthetic agent and it is a ultra-short acting benzodiazepine with a context sensitive half time of 7.5 minutes. Remimazolam is known for its hemodynamic stability compared to propofol. Previous studies have also shown that remimazolam can be safely used in patients with severe aortic stenosis and in cardiac anesthesia induction and during cardiopulmonary bypass. However, there is no definite data on comparison of hemodynamic variables between remimazolam based total intravenous anesthesia (TIVA) and conventional propofol induction and sevoflurane maintenance anesthesia. Therefore, this study is designed to compare effects of remimazolam vs. sevoflurane anesthesia on intraoperative hemodynamics in patients undergoing minimally invasive aortic valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years old
* Patients with severe aortic stenosis, undergoing minimally invasive aortic valve replacement surgery

Exclusion Criteria:

* Patients with known allergy to benzodiazepine, flumazenil, propofol
* Patients with galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Patients with hypersensitivity to Dextran40
* Patients who have been taking benzodiazepine for long term
* Patients with whom heart rate assessment is not accurate, such as atrial fibrillation
* Patients with end stage renal disease requiring hemodialysis
* Patients with history of acute angle glaucoma
* Patients with valve disease severity of grade III or higher, other than aortic valve
* Emergency operation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Total dose of vasopressors and inotropics used. | Start of anesthesia to end of anesthesia
  Total dose of vasopressors and inotropics used during anesthesia will be compared between two groups.

SECONDARY OUTCOMES:
Hypotension and bradycardia event duration | Start of anesthesia to end of anesthesia
  Hypotension and bradycardia event duration will be compared
Extubation time | End of anesthesia to extubation
  Extubation time between the two groups will be compared
Emergence agitation | Arrival of patient at ICU
  Emergence agitation will be compared between the two groups using Riker Sedation-Agitation Scale upon arrival at ICU. The Riker Sedation-Agitation Scale uses a numeric score from 1 (unarousable) to 7 (dangerous agitation)to assess the level of patient sedation and identifies seven levels of sedation and agitation, which range from deep sedation (unarousable) to dangerous agitation.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Study Director — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No